CLINICAL TRIAL: NCT01895543
Title: A Multicenter, Open-label, Safety and Tolerability Extension Trial of 5 mg and 10 mg Elobixibat Daily in the Treatment of Chronic Idiopathic Constipation
Brief Title: Safety and Tolerability Extension Trial for Patients With Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000081; 2012-005601-46 (EudraCT Number)
Record Dates: First submitted 2013-06-28; First posted 2013-07-10 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — elobixibat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EBX10 (Experimental): Elobixibat 10 mg
  Interventions: Drug: Elobixibat 10 mg

INTERVENTIONS:
Drug: Elobixibat 10 mg — 10 mg Elobixibat daily, with possibility for dose adjustment to 5 mg daily.

SUMMARY:
Safety and Tolerability Extension Trial for Patients with Chronic Idiopathic Constipation (CIC)

DETAILED DESCRIPTION:
This was a Phase 3 multicenter, open-label, safety and tolerability extension trial of 10 mg elobixibat daily, with possibility for dose adjustment to 5 mg daily, for 52-week Treatment Period in patients with CIC. A dose adjustment to 5 mg/day was allowed for the remainder of the trial if a patient reported unacceptable treatment-related diarrhoea that occurred within the first four weeks of treatment.

The trial enrolled patients from two lead-in, double-blind efficacy trials (trial codes NCT01827592 and NCT01833065).

ELIGIBILITY:
Inclusion Criteria:

* Has completed double-blind treatment in either of the lead-in efficacy trials, 000079 or 000080.
* The patient reports having understood and has signed the Informed Consent Form (ICF) and is willing to comply with all trial visits and assessments.
* The patient agrees to refrain from making any new, major lifestyle changes that may affect CIC symptoms (i.e., starting a new diet, changing an exercise plan) from the time of signing the ICF through to the last trial visit.

Exclusion Criteria:

* The patient has been withdrawn/discontinued from the 000079 or 000080 trials.
* The patient is not willing to abide by the restrictions for intake of prohibited medication.
* Women of childbearing potential (defined, for the purpose of this trial, as all females post-puberty, not postmenopausal ≥2 years, or not surgically sterile) who have a positive urine pregnancy test at Visit 1, or who do not agree to use one of the following methods of birth control from the day of signing the ICF until 30 days after the final dose of trial drug are excluded:

  1. Transdermal patch
  2. Established use of oral, injected or implanted hormonal methods of contraception
  3. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
  4. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
  5. Male sterilisation (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
  6. True sexual abstinence: when this is in line with the preferred and usual lifestyle of the patient.
* The patients is considered by the Investigator to be unsuitable to participate in the trial for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (62):
- United States (53):
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Skyline Research, LLC, Cerritos, California
  - West Gastroenterology Associates, Los Angeles, California
  - Sacramento Research Medical Group, Sacramento, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Zasa Clinical Research, Boynton Beach, Florida
  - Meridien Research, Bradenton, Florida
  - Pulmonary Associates of Brandon, Brandon, Florida
  - Health Care Family Rehab Corp., Hialeah, Florida
  - Medsearch Professional Group, Inc., Hialeah, Florida
  - The Community Research of South Florida, Hialeah, Florida
  - Center for Gastrointestinal Disorders, Hollywood, Florida
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Jupiter Research Inc., Jupiter, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Research Institute of South Florida, Miami, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Mount Vernon Clinical Research, Atlanta, Georgia
  - Georgia Clinical Research, Snellville, Georgia
  - Evanston Hospital, Evanston, Illinois
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - ActivMed Practices and Research, Inc., Newington, New Hampshire
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Carolina Digestive Health Associates, PA, Concord, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - PharmQuest, LLC, Greensboro, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - TriHealth, Inc., Cincinnati, Ohio
  - Clinical Research Associates, LLC, Oklahoma City, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Family Medical Associates, Levittown, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Anderson Gastroenterology Associates, Anderson, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Memphis Gastroenterology Group, PC, Germantown, Tennessee
  - Associates in Gastroenterology, LLC, Hermitage, Tennessee
  - HCCA Clinical Research Solutions, Jackson, Tennessee
  - KRK Medical Research, Dallas, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Pioneer Research Solutions, Inc., Sugar Land, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Northwest Gastroenterology Associates, Bellevue, Washington
- Cliniques Universitaires Saint Luc (there may be other sites in this country), Brussels, Belgium
- Prime Health Clinical Research Organization (there may be other sites in this country), Toronto, Ontario, Canada
- Gastroenterologie, s. r. o. (there may be other sites in this country), Hradec Králové, Czechia
- Pannónia Magánorvosi Centrum Kft. (there may be other sites in this country), Budapest, Hungary
- SPZOZ Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi (there may be other sites in this country), Lódz, Łódź Voivodeship, Poland
- KM Management sro (there may be other sites in this country), Nitra, Slovakia
- Louise Lelpoldt Medical Centre (there may be other sites in this country), Bellville, Western Cape, South Africa
- Uppsala Akademiska Sjukhus (there may be other sites in this country), Uppsala, Sweden
- Synexus Merseyside Clinical Research Centre (there may be other sites in this country), Liverpool, England, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial enrolled patients from two lead-in, double-blind efficacy trials (000079 and 000080).
Period: Overall Study
Arm/Group | EBX10
Started | 411
Safety Analysis Set | 409 (Set included all enrolled patients who took at least one dose of Investigational Medicinal Product.)
Per Protocol Analysis Set | 380 (Set included all enrolled patients who had no major protocol deviations.)
Completed | 282
Not Completed | 129
Not completed — Withdrawal by Subject | 43
Not completed — Lost to Follow-up | 25
Not completed — Adverse Event | 28
Not completed — Subject's substantial non-compliance | 6
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 2
Not completed — Other (Not fulfilling above criteria) | 24

BASELINE CHARACTERISTICS:
Arm/Group | EBX10
Number analyzed (Participants) | 411
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 362
  >=65 years | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (14.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 351
  Male | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 74
  White | 324
  More than one race | 1
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: Meters (m)] | 1.654 (0.0834)
Weight [Mean (Standard Deviation); unit: Kilogram (Kg)] | 73.61 (14.159)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 26.87 (4.284)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: The Investigator recorded all AEs throughout the trial from the time of obtaining informed consent till the last visit (i.e., Visit 6). Information on AE was collected at each visit. All AEs were recorded in AE log for each patient.
Time Frame: For the overall 52-week Treatment Period
Population: Safety Analysis Set
Measure: Number; unit: Patients
Arm/Group | EBX10
Number analyzed (Participants) | 409
Patients
  AEs | 241
  SAEs | 14

2. Primary Outcome: Incidence of Markedly Abnormal Changes in Clinical Safety Laboratory Variables
Description: Outcome measure include laboratory parameters from haematology, coagulation and clinical chemistry
Time Frame: For the overall 52-week Treatment Period
Population: Safety Analysis Set
Measure: Number; unit: Patients
Arm/Group | EBX10
Number analyzed (Participants) | 409
Patients
  Gamma Glutamyl Transferase (Units/Litre): >3*ULN | 6
  Triglycerides : >3.39 millimoles/Litre | 5
  LDL Cholesterol : >4.1 millimoles/Litre | 3
  Glucose : <2.2 (F) and <2.8 (M) millimoles/Litre | 3
  Activated Partial Thromboplastin Time : >70 second | 3
  Prothrombin Time : >25 seconds | 2
  Sodium : >155 millimoles/Litre | 2
  Chloride : <90 millimoles/Litre | 2
  Alanine Aminotransferase : >3*ULN | 1
  Erythrocytes (10^12/L) : <3.1 | 1
  Potassium : >6.5 millimoles/Litre | 1
  Glucose : >22.2 millimoles/Litre | 1

3. Primary Outcome: Incidence of Markedly Abnormal Changes in Electrocardiograms (ECGs)
Description: A routine 12-lead ECG was performed at all visits. The ECG included heart rate, PR, QRS, and QT intervals assessment.
Time Frame: For the overall 52-week Treatment Period
Population: Safety Analysis Set
Measure: Number; unit: Patients
Arm/Group | EBX10
Number analyzed (Participants) | 409
Patients | 3

4. Primary Outcome: Incidence of Markedly Abnormal Changes in Body Weight and Vital Signs
Description: Vital signs were measured at all visits and included blood pressure (BP: measured after the patient had been in a seated position for ≥3 minutes of rest), pulse, respiration rate, body temperature, and body weight.
Time Frame: For the overall 52-week Treatment Period
Population: Safety Analysis Set
Measure: Number; unit: Patients
Arm/Group | EBX10
Number analyzed (Participants) | 409
Patients
  Temperature - <35^0 celsius | 2
  Diastolic BP - >105 mmHg | 2
  Diastolic BP - <50 mmHg | 1
  Systolic BP - <85 mmHg | 1

5. Secondary Outcome: Use of Concomitant Over-the-counter (OTC) Laxatives
Description: The use of OTC laxatives during the trial was assessed based upon the concomitant medication module of the electronic Case Report Form (eCRF).
Time Frame: For the overall 52-week Treatment Period
Population: Safety Analysis Set
Measure: Number; unit: Patients
Arm/Group | EBX10
Number analyzed (Participants) | 409
Patients
  Contact laxatives | 33
  Osmotically acting laxatives | 14
  Softeners, Emollients | 11
  Bulk Producers | 6
  Enemas | 1

6. Secondary Outcome: Change From Baseline in Global Evaluation of Constipation Severity
Description: The constipation severity score was measured on a 5-point scale (1: none to 5: very severe).
Time Frame: At Week 12, 24, 36, and 52
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | EBX10
Number analyzed (Participants) | 409
Unit on a scale
  At Week 12 | -0.2 (1.10)
  At Week 24 | -0.2 (1.10)
  At Week 36 | -0.1 (1.11)
  At Week 52 | -0.2 (1.08)

7. Secondary Outcome: Change From Baseline in Global Evaluation of Treatment Effectiveness
Description: The treatment effectiveness score was measured on a 5-point scale (1: extremely effective, 2: quite a bit effective, 3: moderately effective, 4: little bit effective, 5: not at all effective).
Time Frame: At Week 12, 24, 36, and 52
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | EBX10
Number analyzed (Participants) | 409
Unit on a scale
  At Week 12 | -0.6 (1.43)
  At Week 24 | -0.6 (1.36)
  At Week 36 | -0.7 (1.24)
  At Week 52 | -0.7 (1.22)

8. Secondary Outcome: Change From Baseline in Patient Assessment of Constipation - Quality of Life (PAC-QOL): Overall Score
Description: PAC-QOL is a 28-item questionnaire for psychometric assessment of disease-specific QOL. The questionnaire is based on a 5-point Likert scale; ranging from 0 [none of the time or not at all] to 4 [all of the time or extremely]). A lower score indicates a better QOL. The PAC-QOL questionnaire is developed specifically for patients with constipation. PAC-QOL has four sub-scales: 'Worries and Concerns', 'Physical Discomfort', 'Psychosocial Discomfort', and 'Dissatisfaction'.
Time Frame: At Week 12, 24, 36 and 52
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | EBX10
Number analyzed (Participants) | 409
Unit on a scale
  At Week 12 | -0.24 (0.677)
  At Week 24 | -0.21 (0.639)
  At Week 36 | -0.16 (0.687)
  At Week 52 | -0.22 (0.644)

9. Primary Outcome: Number of Patients Using Concomitant Medications
Description: The concomitant medications details were collected throughout the trial at all visits. Data were obtained at scheduled or unscheduled trial visits based on information provided spontaneously by the patient or as a result of questioning the patient.
Time Frame: For the overall 52-week Treatment Period
Population: Safety Analysis Set
Measure: Number; unit: Patients
Arm/Group | EBX10
Number analyzed (Participants) | 409
Patients | 340

10. Secondary Outcome: Change From Baseline in EuroQol Group 5-Dimensions 5-Level Questionnaire (EQ-5D-5L) Scores
Description: EQ-5D-5L is a standardised measure of health status developed to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L descriptive system comprises the following five dimensions: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels (1-5 denotes): no problems, slight problems, moderate problems, severe problems, and extreme problems, respectively. A unique health state was defined by combining 1 level from each of the 5 dimensions. Each health state was converted into a single EQ-5D-5L index value. The index values are country specific and values specified for United Kingdom (UK) were used for this study. The index value range for UK lies between -0.594 - 1.000. A positive index value represents better health status while the negative value represents poor health status.
Time Frame: At Week 12, 24, 36 and 52
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | EBX10
Number analyzed (Participants) | 409
Unit on a scale
  At Week 12 | 0.0 (0.14)
  At Week 24 | 0.0 (0.14)
  At Week 36 | 0.0 (0.15)
  At Week 52 | 0.0 (0.15)

11. Secondary Outcome: Change From Baseline in EuroQol Group Visual Analog Scale (EQ-VAS) Score
Description: The EQ VAS presents the participant's self-evaluated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. This scale is numbered from 0 to 100, where '100' means best health you can imagine and '0' means worst health you can imagine. The participant simply mark an 'X' on the scale to indicate "how his/her health is TODAY" and mention the same number in a box provided.
Time Frame: At Week 12, 24, 36 and 52
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | EBX10
Number analyzed (Participants) | 409
Unit on a scale
  At Week 12 | 0.7 (13.43)
  At Week 24 | 1.2 (11.95)
  At Week 36 | 1.0 (12.44)
  At Week 52 | 0.8 (12.35)

ADVERSE EVENTS:
Time Frame: For the overall 52-week Treatment Period and the 2-week Follow-up Period
Description: The Investigator monitored the condition of the patient and recorded all AEs throughout the trial from the time of obtaining informed consent until the last visit (i.e. Visit 6 - the end of the follow-up period) in the AEs Log . Information on AEs was collected at each trial visit.
Groups:
- EBX 10: Elobixibat 10 mg
  Elobixibat 10 mg: 10 mg Elobixibat daily, with possibility for dose adjustment to 5 mg daily.
Arm/Group | EBX 10
Serious Adverse Events (participants affected / at risk) | 14/409
Other Adverse Events (participants affected / at risk) | 77/409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBX 10 (N=409)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2)
Breast abscess (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Emotional distress (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBX 10 (N=409)
Abdominal pain (Gastrointestinal disorders) | 28 (31)
Diarrhoea (Gastrointestinal disorders) | 57 (69)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.